CLINICAL TRIAL: NCT06736860
Title: Early and Precise Application and Evaluation of Tranexamic Acid in Patients With Traumatic Bleeding Based on Dynamic Monitoring of Thromboelastography
Brief Title: Tranexamic Acid in Patients With Traumatic Bleeding Based on Dynamic Monitoring of Thromboelastography
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-615
Record Dates: First submitted 2024-12-06; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Trauma Coagulopathy
Keywords: Trauma Coagulopathy; tranexamic acid; Thromboelastography
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1+1 control group (Active Comparator): Early prehospital administration of TXA 1 g intravenously followed by a continuous infusion of 1 g tranexamic acid (TXA) over 8 hours
  Interventions: Drug: Tranexamic acid (TXA) injection
- 1+X the case group (Experimental): Early prehospital administration of TXA 1 g , then using thromboelastography (TEG) to assess the need for a second or even multiple administrations of TXA ( 1+X regimen) in addition to the administration of 1 g of TXA intravenously
  Interventions: Drug: Tranexamic acid (TXA) injection

INTERVENTIONS:
Drug: Tranexamic acid (TXA) injection — All enrolled patients with acute trauma were given 1 g tranexamic acid (TXA) within 3 h after trauma, which was infused intravenously within 10 min, and randomized into groups. After admission, the first laboratory examination was conducted for both groups. The 1+1 control group continued to infuse 1g TXA within 8 h.
  Arms: 1+1 control group
Drug: Tranexamic acid (TXA) injection — All enrolled patients with acute trauma were given 1 g tranexamic acid (TXA) within 3 h after trauma, which was infused intravenously within 10 min, and randomized into groups. After admission, the first laboratory examination was conducted for both groups. the 1+x study group was subjected to thromboelastography (TEG) without TXA for the time being, and the coagulation and fibrinolytic status of the patients was judged according to the results of TEG (LY30, EPL value), and the patients diagnosed with hyperfibrinolysis continued to be infused with 1g TXA, and the patients diagnosed with normal or reduced fibrinolysis were not infused with TXA. TEG was rechecked after 4 h, and the decision of whether to use TXA was based on the TEG results.
  Arms: 1+X the case group

SUMMARY:
Trauma is an important global public health problem and is the leading cause of death in people under 40 years old. Studies have shown that early prehospital administration of TXA 1 g intravenously followed by a continuous infusion of 1 g tranexamic acid (TXA) over 8 hours ( 1+1 regimen) is effective in reducing mortality in trauma patients, but there is a residual risk of death. This clinical study utilized real-time dynamic monitoring of coagulation fibrinolytic status in trauma patients using thromboelastography (TEG) to assess the need for a second or even multiple administrations of TXA (1+X regimen) in addition to the administration of 1 g of TXA intravenously and to compare the two mortality rates, thus guiding the early and precise use of TXA in trauma patients to potentially reduce mortality in trauma patients while decreasing thromboembolic risk. The present study is an optimization and addition to the TXA 1+1 regimen. Currently, no relevant studies have been reported. This study has important clinical significance for standardizing the early and precise use of TXA in trauma patients and improving the effectiveness and safety of TXA.

DETAILED DESCRIPTION:
Trauma, an important global public health problem, is the leading cause of death in people under 40 years of age. Post-traumatic hemorrhage deaths account for approximately half of the 4.6 million injury deaths worldwide each year . Their early deaths are due to severe hemorrhage and later to traumatic brain injury or secondary multi-organ dysfunction. Although resuscitation protocols for post-traumatic hemorrhage have improved over the past decade, shifting from massive rehydration aimed at perfusion to "damage control resuscitation" that prioritizes correction of early coagulation abnormalities, current transfusion therapies are still unable to correct coagulation during sustained bleeding. In recent years, the hemostatic drug therapy represented by Tranexamic Acid (TXA) has incorporated antifibrinolytic drugs into the global trauma practice guidelines . Overseas studies have shown that the use of TXA within 3 h after trauma can reduce the mortality rate due to trauma bleeding [5,6], but domestic clinical studies in this area are less reported, which is worthy of in-depth study.

The use of TEG for real-time dynamic monitoring of coagulation and fibrinolytic status in trauma patients to guide the early and precise application of TXA may be effective in reducing the mortality rate of severely traumatized patients, as well as reducing the occurrence of thromboembolism. Since the half-life of tranexamic acid is 1.8h , the present study is to use TEG to monitor the coagulation fibrinolytic status of traumatized patients in real time, and to assess the need for secondary or even multiple administrations of TXA (up to three times) (i.e., the 1+X regimen) after two half-life periods of TXA are about to be metabolized on the basis of the intravenous injection of 1g of TXA and to compare the two mortality rates, so that the early and precise use of TXA in traumatized patients can be guided, which may be effective in reducing the occurrence of thromboembolism. patients to guide the early and precise use of TXA in trauma patients, potentially reducing mortality in trauma patients while reducing the risk of thromboembolism. The present study is an optimization and addition to the TXA 1+1 regimen. Currently, there are no relevant literature reports and no references in relevant clinical trial registry websites. This study is clinically important for standardizing the early and precise use of TXA in trauma patients and improving the effectiveness and safety of TXA.

ELIGIBILITY:
Inclusion Criteria:

1. . trauma patients 18 -80 years of age (50 points > trauma ISS score > 16);
2. . hypotension (systolic blood pressure ≤ 90 mm Hg) and/or tachycardia (heart rate ≥ 110 beats/min);
3. . receiving a 1 g TXA push within 3 h of the injury, with the push completed within 10 min of arrival at the hospital.
4. . signing the informed consent form.

Exclusion Criteria:

1. .Coagulation abnormalities due to co-morbid hematologic or autoimmune diseases
2. Inability to establish venous or intraosseous access
3. Pregnant women
4. Traumatic cardiac arrest for more than 5 minutes
5. Failure of cardiopulmonary resuscitation
6. Penetrating brain injury
7. Drowning or hanging -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality rate | 30-day

SECONDARY OUTCOMES:
24-h and hospitalized mortality rates | Day1 and through study completion, an average of 7day
24 h of blood component transfusion | day1
Incidence of multi-organ failure | through study completion, an average of a week
Incidence of thrombotic events during hospitalization | through study completion, an average of a week

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Because the data may be used for multiple analyses and article writing, the data will not be shared at this time.